CLINICAL TRIAL: NCT00667264
Title: Ambulatory Continuous Peripheral Nerve Blocks for Treatment of Post-Amputation Phantom Limb and Stump Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Summit Medical (Unknown); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Associate Professor, In Residence, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCSD Phantom Pilot; GM077026
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Amputation; Phantom Limb; Stump Pain
Keywords: pain; phantom limb; stump pain; catheter; nerve block; peripheral nerve block; ucsd; Post-amputation phantom limb or stump pain
MeSH Terms: conditions — Phantom Limb; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Active Comparator): 3-7 days of perineural local anesthetic infusion
  Interventions: Procedure: perineural ropivacaine
- Placebo (Placebo Comparator): 3-7 days of perineural normal saline infusion
  Interventions: Procedure: perineural ropivacaine

INTERVENTIONS:
Procedure: perineural ropivacaine — Subjects will be randomized to one of two groups: ropivacaine 0.4% or normal saline (placebo). The basal rate will be set at 7 mL/h.

SUMMARY:
Research study to determine if putting local anesthetic-or numbing medication-through one or two tiny tube(s) placed next to the nerves that go to an amputated limb will decrease phantom limb and/or stump pain.

DETAILED DESCRIPTION:
Specific Aim 1: To determine if, compared with current standard-of-care treatment, the addition of an ambulatory continuous peripheral nerve block decreases post-amputation phantom limb and stump pain.

Hypothesis 1: Following upper or lower extremity amputation, phantom limb and/or stump pain will be significantly decreased four weeks following a multiple-day ambulatory continuous peripheral nerve block as compared with patients receiving standard-of-care treatment (as measured on the 11-point numeric rating scale).

Specific Aim 2: To investigate the possible relationship between the addition of a multiple-day ambulatory continuous peripheral nerve block to standard-of-care treatment of post-amputation phantom limb and/or stump pain and cortical reorganization.

Hypothesis 2: Following upper or lower extremity amputation with subsequent phantom limb pain/sensation and/or stump pain, the addition of a multiple-day ambulatory continuous peripheral nerve block to standard-of-care treatment will result in cortical reorganization during and four-weeks following the perineural infusion (as measured by MRI).

ELIGIBILITY:
Inclusion Criteria:

* previous upper or lower limb amputation including at least one metacarpal or metatarsal bone, respectively
* age 18 years or older
* phantom limb and/or stump pain described as at least a 2 on the NRS for the previous week [and pain occurring on a weekly basis over the previous month]
* willing to have an ambulatory perineural infusion for 6 days
* willing to avoid additional "new" analgesic interventions from 4 weeks prior to at least 4 weeks following catheter placement, and preferably to 6 months following catheter placement
* the availability of a "caretaker" who will transport the subject home following the procedure and remain with the subject for the first night of the infusion

Exclusion Criteria:

* known hepatic or renal insufficiency
* allergy to the study medications
* possessing a contraindication to perineural catheter placement or perineural local anesthetic infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-10; Primary Completion 2011-01 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Primary analysis will compare the two treatment groups for the phantom limb/stump pain change from baseline to 4 weeks following the initial catheter placement | Week 4

SECONDARY OUTCOMES:
Physical Functioning · Brief Pain Inventory | pre-intervention, then days 1, 3, 8, 28, 84, and 365
Nervous System Reorganization [if patient elected to participate in the MRI procedures] · MRI procedure | pre-intervention; and then 8 and 28 days post-intervention
Pain · 11-point numeric rating scale of pain intensity · Usage of baseline and rescue analgesics in previous 24 hours · Patient Global Impression of Change scale | Day 8, Day 28, Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Brian Ilfeld, M.D., M.S., Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Medical Center, San Diego, California, United States